CLINICAL TRIAL: NCT00813228
Title: Assessment of the Effects of a DPP-4 Inhibitor (Sitagliptin) Januvia on Immune Function in Healthy Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 090055; 09-DK-0055
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11-26

CONDITIONS: Diabetes Mellitus Type 1; Diabetes Mellitus Type 2
Keywords: Immune Function; DDP-4; Sitagliptin; GLP-1; TGF Beta
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Camurati-Engelmann Syndrome | interventions — Sitagliptin Phosphate

INTERVENTIONS:
Drug: Sitagliptin (Januvia)

SUMMARY:
Patients with diabetes have high blood sugar levels (hyperglycemia) because pancreatic beta-cells no longer produce sufficient insulin. Insufficient beta-cell function can be caused by an autoimmune killing of the beta-cells in type 1 diabetes (T1D), or by poorly understood mechanisms in type 2 diabetes (T2D). Glucagon-like peptide-1 (GLP-1) improves function of the insulin-producing beta cells, but GLP-1 has a very short circulating half-life because it is cleaved by the enzyme dipeptidyl peptidase IV (DPP-4). One current treatment being used to improve glycemia control in patients with T2D is sitagliptin, an inhibitor of DPP-4. By inhibiting DPP-4, sitagliptin increases GLP-1 levels, resulting in improved beta cell function. Sitagliptin is now being tested in individuals with new-onset T1D to determine whether it may help to preserve beta cell function. Because T1D is a disease in which the immune system destroys the insulin-producing beta cells in the pancreas, we wish to determine if and how sitagliptin alters immune function. Sitagliptin has been shown by Merck to be safe and effective with no overt immuno-toxicities. However, several lines of evidence suggest that DPP-4 inhibitors such as sitagliptin could be immunomodulatory.

This randomized clinical trial will study immune function in healthy volunteers given short-term (4 week) treatment with either sitagliptin or placebo. During the study, we will take blood samples at various time intervals before, during and after treatment. We will compare the immune response with and without sitagliptin treatment using blood samples from healthy individuals. We will measure changes in the magnitude and type of immune responses. The study period is nine weeks. The study s primary outcome will be changes in blood plasma levels of a protein marker associated with decreased inflammation: Transforming Growth Factor Beta 1 (TGF beta 1). In addition, we plan to use these blood samples to measure sitagliptin s effect on expression levels of several cytokines (immune proteins). We will also measure the level of proliferation in stimulated PBMCs (blood immune cells) and gene expression in whole blood after sitagliptin treatment.

DETAILED DESCRIPTION:
Patients with diabetes have high blood sugar levels (hyperglycemia) because pancreatic b-cells no longer produce sufficient insulin. Insufficient b-cell function can be caused by an autoimmune killing of the b-cells in type 1 diabetes (T1D), or by poorly understood mechanisms in type 2 diabetes (T2D). Glucagon-like peptide -1 (GLP-1) improves function of the insulin-producing beta cells, but GLP-1 has a very short circulating half-life because it is cleaved by the enzyme dipeptidyl peptidase IV (DPP-4). One current treatment being used to improve glycemia control in patients with T2D is sitagliptin, an inhibitor of DPP-4. By inhibiting DPP-4, sitagliptin increases GLP-1 levels resulting in improved beta cell function. Sitagliptin is now being tested in individuals with new-onset T1D to determine whether it may help to preserve beta cell function. Because T1D is a disease in which the immune system destroys the insulin-producing beta cells in the pancreas, we wish to determine if and how sitagliptin alters immune function. Sitagliptin has been shown by Merck to be safe and effective with no overt immuno-toxicities. However, several lines of evidence suggest that DPP-4 inhibitors such as sitagliptin could be immunomodulatory.

This randomized clinical trial will study immune function in healthy volunteers given short-term (4 week) treatment with either sitagliptin or placebo. During the study, we will take blood samples at various time intervals before, during and after treatment. We will compare the immune response with and without sitagliptin treatment using blood samples from healthy individuals. We will measure changes in the magnitude and type of immune responses. The study period is nine weeks. The study s primary outcome will be changes in blood plasma levels of a protein marker associated with decreased inflammation: Transforming Growth Factor-Beta1 (TGFb1). In addition, we plan to use these blood samples to measure sitagliptin s effect on expression levels of several cytokines (immune proteins). We will also measure the level of proliferation in stimulated PBMCs (blood immune cells) and gene expression in whole blood after sitagliptin treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age greater than 18

Fasting blood glucose less than 100 mg/dl, and a normal Hgb A1c (less than 5.7%),

Available for follow up through 9 weeks.

In good general health without clinically significant medical history as deemed by study investigators.

EXCLUSION CRITERIA:

History of diabetes or other autoimmune diseases including (but not limited to) rheumatoid arthritis, lupus, multiple sclerosis.

Active hepatitis B, C and/ or HIV infection.

Recent diagnosis or active treatment for malignancy.

Recent (within 3 weeks) severe allergy symptoms such as allergy-induced asthma, skin eruptions or urticaria.

Recent (within 3 weeks) viral or bacterial infections.

History of other immune abnormalities, or the presence of disease processes or medications that, in the opinion of the investigator, may alter immune function.

Pregnant and nursing females.

Women who have child-bearing potential but not using adequate birth control.

History of hypersensitivity reaction to sitagliptin.

History of anemia (based on the NIH laboratory department hemoglobin reference range for normal individuals).

History of pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-01-06; Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Changes in plasma TGF-Beta 1 levels.

SECONDARY OUTCOMES:
Changes in plasma or stimulated PBMC cytokines levels, changes in stimulated PBMC proliferation, changes in peripheral blood gene expression and changes in immune phenotyping.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina I Rother, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Drucker DJ. Glucagon-like peptide-1 and the islet beta-cell: augmentation of cell proliferation and inhibition of apoptosis. Endocrinology. 2003 Dec;144(12):5145-8. doi: 10.1210/en.2003-1147. No abstract available. PMID 14645210
- [Background] Thompson MA, Ohnuma K, Abe M, Morimoto C, Dang NH. CD26/dipeptidyl peptidase IV as a novel therapeutic target for cancer and immune disorders. Mini Rev Med Chem. 2007 Mar;7(3):253-73. doi: 10.2174/138955707780059853. PMID 17346218
- [Background] Amori RE, Lau J, Pittas AG. Efficacy and safety of incretin therapy in type 2 diabetes: systematic review and meta-analysis. JAMA. 2007 Jul 11;298(2):194-206. doi: 10.1001/jama.298.2.194. PMID 17622601